CLINICAL TRIAL: NCT05523635
Title: Post Market Clinical Evaluation of Gamma 4: Prospective, Multicenter, Follow-up Study (PEGASUS)
Brief Title: Post Market Clinical Evaluation of Gamma 4
Acronym: PEGASUS
Status: Active, not recruiting | Type: Observational
Sponsor: Stryker Trauma and Extremities (Industry)
Responsible Party: Sponsor
Other Study IDs: TA-01-2022
Record Dates: First submitted 2022-08-04; First posted 2022-08-31 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Femoral Fracture
Keywords: Fractures; Hip Fracture; Leg Injuries; Wounds and Injuries
MeSH Terms: conditions — Femoral Fractures; Fractures, Bone; Hip Fractures; Leg Injuries; Wounds and Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Gamma 4: Subjects in the clinical investigation will undergo placement of the Gamma4 Nailing System, according to the approved Instructions for Use and Operative Technique Manual
  Interventions: Device: Gamma4 Nailing System

INTERVENTIONS:
Device: Gamma4 Nailing System — The Gamma4 Nailing System is is indicated for the treatment of stable and unstable fractures as well as for stabilization of bones and correction of bone deformities in the intracapsular, trochanteric, subtrochanteric and shaft regions of the femur (including osteoporotic and osteopenic bone).

SUMMARY:
This is a prospective, multi-center, non-randomized, post-market clinical investigation of the Gamma 4 System. Neither subjects nor investigators are blinded to treatment.

It is anticipated that a total of 100 subjects will be enrolled at five sites. Total duration of enrollment, 12 month follow-up and analysis is expected to take approximately 30 months. The clinical investigation has been designed to follow the surgeon's standard of care for subjects treated with a cephalomedullary nail for femoral fractures or and deformities, in addition to a 12 month follow-up visit.

The primary endpoint of this clinical investigation is demonstration of bone consolidation by 12 months.

DETAILED DESCRIPTION:
The objective of this clinical investigation is to demonstrate the safety and efficacy/performance of the Gamma 4 System. Enrolled subjects will undergo an initial assessment, with follow-up evaluations at 3 Months, 6 Months, and 12 Months after the index procedure.

The primary endpoint of this clinical investigation is demonstration of bone consolidation by 12 months, as measured by the Investigator.

Secondary endpoints will include safety through reporting the incidence of device related intra-operative and post-operative adverse events by 12 months, patient reported outcome measures (SF-35v2 and Modified Harris Hip Score), and other specific health outcomes.

Efficacy will be assessed through non-inferiority of bone consolidation proportion compared to the pooled literature control, as well as the SF-36 score results by 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Subject is a male or non-pregnant female age 18 years or older at the time of surgery;
* Subject is willing and able to give written informed consent and comply with the requirements of this Clinical Investigation Plan; and
* Subject has or is intended to be treated with the Gamma 4 System in accordance with its legally approved Indication for Use (IFU).

Indication For Use in the United States and Canada:

The Gamma4 System is indicated for the treatment of stable and unstable fractures as well as for stabilization of bones and correction of bone deformities in the intracapsular, trochanteric, subtrochanteric and shaft regions of the femur (including osteoporotic and osteopenic bone).

Exclusion Criteria:

* Subject is currently enrolled in or plans to enroll in any concurrent drug and/or device clinical investigation that, in the opinion of the Investigator, may confound results
* Subject with exclusion criteria required by local law
* Subject who is, or will be, inaccessible for follow-up
* Per the Investigator, the subject is in poor general health or undergoing any concurrent disease that would place the subject in excessive risk to surgery (i.e., significant circulatory problems, cardiac disease).
* Any active or suspected latent infection or marked local inflammation in or about the affected area
* Compromised vascularity that would inhibit adequate blood supply to the fracture or the operative site
* Bone stock compromised by disease, infection or prior implantation that cannot provide adequate support and/or fixation of the devices
* Material sensitivity, documented or suspected
* Patients having inadequate tissue coverage over the operative site
* Implant utilization that would interfere with anatomical structures or physiological performance
* Any mental or neuromuscular disorder which would create an unacceptable risk of fixation failure or complications in postoperative care
* Other medical or surgical conditions which would preclude the potential benefit of surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Approximately 100 subjects are to be enrolled in this clinical investigation. Subjects participating in this clinical investigation will be recruited from the investigator's standard subject population, where all subjects presenting for treatment of femoral fractures and deformities with a cephalomedullary nail will be evaluated for clinical investigation participation based on the eligibility criteria.
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2023-03-06 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Bone Consolidation via Clinical Assessment | by 12 months
  Clinical consolidation is defined as no pain or tenderness when weight bearing
Bone Consolidation via Radiographic Assessment | by 12 months
  Radiographic bony consolidation is defined as bridging of the fracture at three of four cortices.

SECONDARY OUTCOMES:
Safety will be measured by capturing the incidence rate of device-related adverse events | 12 months
  Incidence of device related intra-operative and post-operative Adverse Events/incidents by 12 months.
SF-36v2® Physical Component Score and Mental Component Score (PCS & MCS) | 12 months
  The SF-36 PCS is a self-report measure of health status. SF-36 Physical Component Summary scores range from 0 to 100; higher SF-36 score results are linked to better subject results.
  Efficacy/performance at 12 months will be measured by the SF-36 Physical Component Score (PCS) compared to the pooled literature controls.
Modified Harris Hip Score | 12 months
  The modified Harris Hip Score is a hip-specific questionnaire which evaluates hip pain and function. It is a commonly used and validated tool.
  Efficacy/performance at 12 months will be measured by the modified Harris Hip Score compared to the pooled literature controls.

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Gibson, Study Director — Stryker Trauma and Extremities
Locations (5):
- United States (5):
  - William Beaumont Hospital, Royal Oak, Michigan
  - MetroHealth, Cleveland, Ohio
  - UT Health, San Antonio, Texas
  - Inova Health Care Services, Falls Church, Virginia
  - SSM Health - Madison, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No